CLINICAL TRIAL: NCT04769583
Title: A Double Blind Randomized Study for Treatment of Helicobacter Pylori Infection: 14-day Non-bismuth Quadruple Therapy Versus Triple Therapy.
Brief Title: 14-day Quadruple Therapy Versus Triple Therapy in HP Eradication
Acronym: HEPRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: mohamed bouchoucha (Industry)
Responsible Party: Sponsor-Investigator, mohamed bouchoucha, Assistant Clinical Data management, Les Laboratoires des Médicaments Stériles
Organization: Les Laboratoires des Médicaments Stériles (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN2018-INT-INS-14
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Gastritis H Pylori
Keywords: Breath Tests; Helicobacter pylori

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: a placebo which has the same visual characteristics as metronidazole in the boxes of the triple therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concomitant quadruple therapy (QC) (Active Comparator): PPI (esomeprazole: 40 mg x 2 per day) with the amoxicillin (1 g x 2 per day), metronidazole (500 mg x 2 per day) and clarithromycin (500 mg x 2 per day) for 14 days
  Interventions: Drug: metronidazole based quadriple therapy
- triple therapy (TT) (Placebo Comparator): PPI (esomeprazole: 40 mg x 2 per day) with amoxicillin (1 g x 2 per day) and clarithromycin (500 mg x 2 per day) AND PLACEBO for 14 days.
  Interventions: Drug: placebo based quadriple therapy

INTERVENTIONS:
Drug: metronidazole based quadriple therapy — patient randomized in QC will be treated by a double dose PPI (esomeprazole: 40 mg x 2 per day) in combination with amoxicillin (1 g x 2 per day), metronidazole (500 mg x 2 per day) and clarithromycin (500 mg x 2 per day)
  Other Names: concomitant quadruple therapy (QC)
  Arms: concomitant quadruple therapy (QC)
Drug: placebo based quadriple therapy — patient randomized in TT will be treated by double dose PPI (esomeprazole: 40 mg x 2 per day) in combination with amoxicillin (1 g x 2 per day), clarithromycin (500 mg x 2 per day) and a placebo of metronidazole.
  Other Names: Triple therapy (TT)
  Arms: triple therapy (TT)

SUMMARY:
In this prospective randomized-controlled study, treatment-naive H. pylori-infected patients are randomized to receive either standard triple therapy or sequential therapy. The aim is to compare the efficacy of concomitant quadruple therapy with standard triple therapy as a first line treatment for H. pylori infection in Tunisian patients.

DETAILED DESCRIPTION:
This study includes male and female patients aged between 18 and 65, with documented Hp infection and who have had no previous eradication treatment.The diagnosis of Hp infection was made through an anatomopathological study. Gastric biopsies were taken according to the Sydney protocol: two fundics in one pot, two antrals and one at the angle of the lesser curve in a second pot. The biopsies were studied by an experienced anatomopathologist.

The included patients were randomly divided into two treatment groups according to a 1: 1 ratio: the first group received concomitant quadruple therapy (QC) combining a double dose PPI (esomeprazole: 40 mg x 2 per day) with the amoxicillin (1 g x 2 per day), metronidazole (500 mg x 2 per day) and clarithromycin (500 mg x 2 per day) for 14 days. The second group received triple therapy (TT) combining a double dose PPI (esomeprazole: 40 mg x 2 per day) with amoxicillin (1 g x 2 per day) and clarithromycin (500 mg x 2 per day) for 14 days.

H. pylori eradication was assessed by the 13C-urea breath test 8 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 65, with documented Hp infection.

Exclusion Criteria: are excluded patients:

* With Cirrhosis.
* With Renal failure (serum creatinine> 120 µmol / L).
* Having complicated peptic ulcer (stenosis or hemorrhage or perforation) in an acute phase.
* Having severe psychiatric disorders.
* Having had gastric surgery in their history.
* Having already received an HP eradication treatment.
* Having received an antibiotic within the last two weeks.
* Who are allergic to one of the antibiotics used in the anti-Hp cure.
* Who are drug addicted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
HP eradiction rate | 6 weeks after completion of study treatment
  assessment by breath test

SECONDARY OUTCOMES:
percentage of adverse reactions | 3 months
  we will determinate the percentage of adverse reactions in each group of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fattouma Bourguiba Hospital, Monastir, Tunisia